CLINICAL TRIAL: NCT06881290
Title: Pilot Study on the Treatment of Vunakizumab in Mild to Moderate Systemic Lupus Erythematosus
Brief Title: Vunakizumab for the Treatment of Mild to Moderate Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese SLE Treatment And Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTAR011
Record Dates: First submitted 2025-03-10; First posted 2025-03-18 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Vunakizumab; Systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vunakizumab (Experimental)
  Interventions: Drug: Vunakizumab (IL-17A inhibitor)

INTERVENTIONS:
Drug: Vunakizumab (IL-17A inhibitor) — Vunakizumab combined with glucocorticoid therapy: Vunakizumab is administered subcutaneously at 240 mg at weeks 0, 2, and 4, followed by maintenance dosing every 4 weeks at 240 mg per dose.

SUMMARY:
Systemic lupus erythematosus (SLE) is a systemic autoimmune disease characterized by heterogeneous clinical manifestations ranging from mild cutaneous involvement to severe multi-organ damage. While its pathogenesis involves complex cytokine dysregulation, emerging evidence implicates IL-17 as a potential contributor. Elevated serum IL-17 levels have been observed in SLE patients compared to healthy controls, with heightened expression detected in renal and cutaneous lesions. Ustekinumab, a monoclonal antibody targeting IL-23/IL-12 that indirectly modulates IL-17 signaling, demonstrated superior efficacy and safety to placebo in an SLE clinical trial, particularly in glucocorticoid dose reduction. Notably, no clinical trials have directly evaluated IL-17-targeted therapies for SLE, though case reports suggest secukinumab (an anti-IL-17A agent) may improve cutaneous manifestations in psoriasis-SLE overlap patients.

Vunakizumab, a humanized anti-IL-17A monoclonal antibody (IgG1/κ) with a unique epitope-binding profile, selectively inhibits IL-17A-mediated inflammatory signaling. Its established safety profile and infrequent dosing regimen in IL-17-mediated diseases (e.g., psoriasis, psoriatic arthritis) warrant investigation in SLE. The investigators aim to provide new treatment options for SLE patients

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-65 years meeting the 2019 EULAR/ACR classification criteria for SLE.
2. SLEDAI score was within 2-12 scores (with clinical SLEDAI [cSLEDAI] ≠ 0).
3. Occurence of new or recurrent mucocutaneous or joint involvement.
4. Stable standard treatment regimen prior to study entry but not effect: Prednisone or equivalent corticosteroid dose ≤ 20 mg per day for more than 4 weeks; Immunosuppressant less than 1 type for more than 12 weeks, including methotrexate ≤15 mg per week, azathioprine ≤100mg per day, mycophenolate mofetil ≤1.5 g per day, tacrolimus ≤2 mg per day, cyclosporine ≤150 mg per day). Antimalarials was permitted.
5. Body mass index (BMI) 18-35 kg/m² at screening.
6. Clinically eligible for Vunakizumab combination therapy with corticosteroids after investigator assessment.
7. Willing to provide written informed consent with demonstrated compliance.

Exclusion Criteria:

1. SLE with major organ dysfunction including Encephalopathy/cognitive impairment, Renal insufficiency, Cardiac insufficiency (NYHA class III-IV), Pulmonary hypertension/interstitial lung disease
2. Active SLE-related organ involvement: Lupus cerebritis, Active lupus nephritis (proteinuria ≥1g/24h), Myocardial involvement, Gastrointestinal vasculitis, Diffuse alveolar hemorrhage, Thrombocytopenic purpura, Hemophagocytic syndrome, Retinopathy
3. Concurrent autoimmune diseases affecting efficacy assessment (e.g., rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis).
4. Liver dysfunction: ALT/AST >1.5×ULN or total bilirubin >1×ULN.
5. Active malignancy within 5 years or history of malignancy.
6. Comorbidities requiring corticosteroids (e.g., asthma, Crohn's disease).
7. Active infections requiring treatment:Tuberculosis, HBV/HCV/HIV/CMV infections
8. Major surgery within 3 months prior to screening.
9. Hypersensitivity or intolerance to funakizumab.
10. Pregnancy, lactation, or planned pregnancy.
11. Biologic therapy within 3 months (anti-CD20 agents, belimumab, TNF-α inhibitors).
12. Recent intensive therapies: Systemic corticosteroids within 3 months/ Plasmapheresis/IVIG/cyclophosphamide within 3 months
13. Any condition deemed by investigators to compromise study completion or patient safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
the percentage of patients achieving an BICLA response at the end of 24 weeks | From enrollment to the end of treatment at 24 weeks
  The BICLA response was defined as a reduction of all severe (BILAG-2004 A) or moderately severe (BILAG-2004 B) disease activity at baseline to lower levels (BILAG-2004 B, C, or D and C or D, respectively) and no worsening in other organ systems (with worsening defined as ≥1 new BILAG-2004 A item or ≥2 new BILAG-2004 B items); no worsening in disease activity, as determined by the SLEDAI-2K score (no increase from baseline) and by the PGA score (no increase of ≥0.3 points from baseline)

SECONDARY OUTCOMES:
the percentage of patients achieving an BICLA response at the end of 12 weeks | From enrollment to the end of treatment at 12 weeks
  The BICLA response was defined as a reduction of all severe (BILAG-2004 A) or moderately severe (BILAG-2004 B) disease activity at baseline to lower levels (BILAG-2004 B, C, or D and C or D, respectively) and no worsening in other organ systems (with worsening defined as ≥1 new BILAG-2004 A item or ≥2 new BILAG-2004 B items); no worsening in disease activity, as determined by the SLEDAI-2K score (no increase from baseline) and by the PGA score (no increase of ≥0.3 points from baseline)
the percentage of patients achieving SRI-4 response at the end of 24 weeks. | From enrollment to the end of treatment at 24 weeks
  The SRI-4 (SLE Responder Index-4) response was defined as a reduction of at least 4 points in SLEDAI score compared with the baseline level, no new British Isles Lupus Assessment Group (BILAG) A organ domain score or no more than one new BILAG B organ domain score, and no worsening in the Physician's Global Assessment (PGA) (<0.3 points worsening from the baseline level).
the percentage of patients achieving SRI-4 response at the end of 12 weeks. | From enrollment to the end of treatment at 12 weeks
  The SRI-4（SLE Responder Index-4） response was defined as a reduction of at least 4 points in SLEDAI score compared with the baseline level, no new British Isles Lupus Assessment Group (BILAG) A organ domain score or no more than one new BILAG B organ domain score, and no worsening in the Physician's Global Assessment (PGA) (<0.3 points worsening from the baseline level).
Changes from baseline in SLEDAI at 24 weeks | From enrollment to the end of treatment at 24 weeks
  SLEDAI stands for Systemic Lupus Erythematosus Disease Activity Index, with a score of 0-6 representing mild disease activity, 7-12 representing moderate disease activity, and 12-16 representing severe disease activity
Changes from baseline in CLASI at 24 weeks. | From enrollment to the end of treatment at 24 weeks
  CLASI stands for Cutaneous Lupus Erythematosus Disease Area and Severity Index. It is a measure of the severity of skin disease, with scores ranging from 0 to 70, with higher scores indicating more severe disease activity
Changes from baseline in PGA at 24 weeks | From enrollment to the end of treatment at 24 weeks
  PGA stands for Physician's Global Assessment (PGA ) . It is used to assess the activity of systemic lupus erythematosus on a scale ranging from 0 to 3, where 0 indicates no disease activity and 3 indicates the most severe disease activity.
Changes from baseline of the SJC and TJC at 24 weeks | From enrollment to the end of treatment at 24 weeks
  Swollen Joint Count(SJC) and Tender Joint Count(TJC) indicate the number of swollen and tender joints in 28 joints, respectively. 28 joints refer to both shoulders, both elbows, both wrists, both knees, 10 metacarpophalangeal joints, and 10 proximal interphalangeal joints, which ranging from 0 to 28, the higher value means more serious disease activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China